CLINICAL TRIAL: NCT02019771
Title: Prevalence of Gonorrhea and Chlamydia Infections in Multiple Anatomical Sites in HIV-infected Men Who Have Sex With Men at an HIV Clinic in Omaha, Nebraska
Brief Title: Gonorrhea and Chlamydia HIV-infected Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0025-14-FB
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: HIV Infection; Chlamydia; Gonorrhea
Keywords: HIV Infection; Men who have sex with men; Chlamydia; Gonorrhea
MeSH Terms: conditions — HIV Infections; Chlamydia Infections; Gonorrhea; Homosexuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will estimate the rates of asymptomatic Chlamydia and/or Gonorrhea in the oropharynx, rectum and urethra (urine) of HIV infected men who have sex with men at a specialty care center and compare it to the rates in Douglas County, using nucleic acid amplification tests.

DETAILED DESCRIPTION:
Hypothesis: Men who have sex with men (MSM) are at higher risk for sexually transmitted diseases. Currently, free testing for sexually transmitted diseases is only being performed in urine samples. Investigators hypothesize that the rates of both gonorrhea and chlamydia will be higher when testing includes more than one anatomical site (rectum and oropharynx).

The aim of the study is to estimate the rates of asymptomatic Chlamydia and/or Gonorrhea in the oropharynx, rectum and urethra (urine) of HIV infected men who have sex with men at the specialty care center of the University of Nebraska Medical Center and compare to the rates in Douglas County, using nucleic acid amplification tests.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Men with history of sex with men (including transgender and bisexual)
* Older than 19 years of age
* Asymptomatic at the time of visit.

Exclusion Criteria:

* Active sexually transmitted disease symptoms in the oropharynx.
* Recent treatment for Chlamydia or gonorrhea within 3 weeks.
* Treatment with antibiotics active for Chlamydia or gonorrhea within the last 2 weeks: doxycycline, quinolones and azithromycin, and cefixime.
* Women.
* Inability to complete the questionnaire in English or Spanish.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study will be conducted at the Specialty Care Center of the University of Nebraska Medical Center, in Omaha, Nebraska. Adult men who have a history of sex with men who visit the clinic for their appointments will be eligible to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Chlamydia or gonorrhea infection | one day
  Investigators will use nucleic acid amplification tests in urine, rectal and oropharyngeal swab specimens to detect asymptomatic chlamydia and/or gonorrhea infection

SECONDARY OUTCOMES:
accuracy for detecting infection when using one versus 2 versus 3 anatomical sites | 1 day
  Investigators will compare the proportion of infections detected by using only urine, only rectum, only oropharynx vs. using combined sites (urine and rectum, urine and oropharynx or oropharynx and rectum) vs. using all 3 sites.

CONTACTS AND LOCATIONS:
Overall Officials: Uriel S Sandkovsky, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Specialty Care Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Koedijk FD, van Bergen JE, Dukers-Muijrers NH, van Leeuwen AP, Hoebe CJ, van der Sande MA; Dutch STI centres. The value of testing multiple anatomic sites for gonorrhoea and chlamydia in sexually transmitted infection centres in the Netherlands, 2006-2010. Int J STD AIDS. 2012 Sep;23(9):626-31. doi: 10.1258/ijsa.2012.011378. PMID 23033514
- [Result] Bachmann LH, Johnson RE, Cheng H, Markowitz L, Papp JR, Palella FJ Jr, Hook EW 3rd. Nucleic acid amplification tests for diagnosis of Neisseria gonorrhoeae and Chlamydia trachomatis rectal infections. J Clin Microbiol. 2010 May;48(5):1827-32. doi: 10.1128/JCM.02398-09. Epub 2010 Mar 24. PMID 20335410
- [Result] Baker J, Plankey M, Josayma Y, Elion R, Chiliade P, Shahkolahi A, Menna M, Miniter K, Slack R, Yang Y, Masterman B, Margolick JB. The prevalence of rectal, urethral, and pharyngeal Neisseria gonorrheae and Chlamydia trachomatis among asymptomatic men who have sex with men in a prospective cohort in Washington, D.C. AIDS Patient Care STDS. 2009 Aug;23(8):585-8. doi: 10.1089/apc.2008.0277. No abstract available. PMID 19591608
- [Result] Hoover KW, Butler M, Workowski K, Carpio F, Follansbee S, Gratzer B, Hare B, Johnston B, Theodore JL, Wohlfeiler M, Tao G, Brooks JT, Chorba T, Irwin K, Kent CK; Evaluation Group for Adherence to STD and Hepatitis Screening. STD screening of HIV-infected MSM in HIV clinics. Sex Transm Dis. 2010 Dec;37(12):771-6. doi: 10.1097/OLQ.0b013e3181e50058. PMID 20585275
- [Result] Kent CK, Chaw JK, Wong W, Liska S, Gibson S, Hubbard G, Klausner JD. Prevalence of rectal, urethral, and pharyngeal chlamydia and gonorrhea detected in 2 clinical settings among men who have sex with men: San Francisco, California, 2003. Clin Infect Dis. 2005 Jul 1;41(1):67-74. doi: 10.1086/430704. Epub 2005 May 26. PMID 15937765
- [Result] Morris SR, Klausner JD, Buchbinder SP, Wheeler SL, Koblin B, Coates T, Chesney M, Colfax GN. Prevalence and incidence of pharyngeal gonorrhea in a longitudinal sample of men who have sex with men: the EXPLORE study. Clin Infect Dis. 2006 Nov 15;43(10):1284-9. doi: 10.1086/508460. Epub 2006 Oct 10. PMID 17051493